CLINICAL TRIAL: NCT02678039
Title: Fluoroscopy-guided Versus Traditional Placement of Epidural Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPHS#23226
Record Dates: First submitted 2016-01-20; First posted 2016-02-09 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Pain, Postoperative; Pain, Chronic
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Fluoroscopy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoroscopy (Experimental): Real-time fluoroscopic X-ray guidance to confirm placement of an epidural catheter in the spinal epidural space at the desired location.
  Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr into the epidural catheter during and after surgery for pain control.
  Interventions: Device: Fluoroscopy
- Traditional (Active Comparator): The traditional approach for placement of an epidural catheter is used with indirect indicators of placement including palpation of spine and 'loss-of-resistance' to fluid injection.
  Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr into the epidural catheter during and after surgery for pain control.
  Interventions: Procedure: Traditional

INTERVENTIONS:
Device: Fluoroscopy — Device: Fluoroscopy Patients lie prone on X-ray compatible operating table and an X-ray device obtains X-ray images of epidural catheter placement. An epidural catheter is placed with local anesthesia as a needle that is advanced into the epidural space. A catheter is then placed through the needle to the desired location and the needle is removed. After the catheter is placed, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected into the catheter to exclude intravascular placement. Following this, a continuous infusion of 1/8% bupivacaine is started at 4ml/hr. After surgery, the bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusion rate by 2ml/hr up to a maximum of 14ml/hr
  Arms: Fluoroscopy
Procedure: Traditional — An epidural catheter is placed before surgery with the patient sitting at bedside. The catheter is placed with local anesthesia using indirect indicators of proper placement: depth of needle insertion and ability to inject solution through the needle ('loss of resistance'). After needle placement in the epidural space, an epidural catheter is threaded through the needle 3-4 cm and the needle removed. After catheter is placement, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected into the catheter to exclude intravascular placement. Following this, a continuous infusion of 1/8% bupivacaine is started at 4ml/hr. After surgery, the bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusion rate by 2ml/hr up to a maximum of 14ml/hr.
  Other Names: Loss of resistance
  Arms: Traditional

SUMMARY:
This is a prospective, randomized, controlled, and single blinded study. All work performed at Dartmouth-Hitchcock Medical Center, a tertiary care and level one trauma center for the state of New Hampshire with 28 operative suites. 100 patients scheduled to undergo thoracotomies are randomized to receive an epidural placed (for postoperative pain control) using either a traditional approach by feeling the spine for landmarks or using fluoroscopic X-ray guidance. Randomization is blinded to both the anesthesia team caring for the patient in the operating room and to one member of the acute pain team who follows the patient after surgery and is responsible for evaluating post operative pain control (dermatomal distribution of sensory blockade and visual analog scale) and pulmonary function (incentive spirometer use). All patients receive a standardized epidural infusion with local anesthetic and additional pain medications as needed.

DETAILED DESCRIPTION:
All epidurals catheters are placed by the Acute Pain Service in the preoperative period in an operating room equipped for fluoroscopy. Patients will have been previously randomized (following written informed consent) to either standard placement of epidural catheters or fluoroscopically-guided placement.

Standard placement (Comparator): According to usual practice, epidurals placed using the standard technique will be placed in the sitting position using a 'loss of resistance' technique. This technique involves approximation of the T7 vertebral body through palpation of the distal aspect of the scapula and identification of midline through palpation of the spinous processes. The skin is then anesthetized with 1% Lidocaine and an 18 gauge Tuohy needle is inserted until there is engagement with the supraspinous and interspinous ligaments. A glass syringe filled with saline and air is then attached to the Tuohy needle, which is slowly advanced until the epidural space is identified with loss of resistance to injection in the glass syringe. The glass syringe is then detached from the Tuohy needle and the epidural catheter is threaded approximately 3-4 cm into the epidural space. The catheter will then be aspirated using a 3ml syringe to confirm that it has not been place in the intravascular or intrathecal space. Five ml of radiopaque dye (omnipaque) will be injected and a single image taken and stored on disc but not read by a clinician. A test dose of 3ml of 1.5% Lidocaine with epinephrine will then be injected to ensure that the catheter is not intravascular.

Fluoroscopically guided epidural placement (Experimental): Patients will be placed in the prone position. Identification of an appropriate interspace (T7-T12) and midline orientation will be accomplished using fluoroscopic guidance. The skin will then be anesthetized and the epidural space identified using the loss of resistance as described above. Fluoroscopy will be used during identification of the epidural space to confirm midline orientation during advancement of the Tuohy needle. Once the epidural space is identified, the epidural catheter will be advanced to the T4 level. The catheter will then be aspirated as above. 5cc of Omnipaque will be injected into the catheter with anterior-posterior and lateral imaging to ensure expected spread of the dye as confirmation of correct placement in the epidural space. The catheter will then be bolused with 3cc of 1.5% lidocaine with epinephrine to ensure that the catheters are not placed intravascularly.

Following epidural placement via either technique, patients will then be transferred to the surgical operating room where an infusion of 1/8% Bupivicaine will be started at a rate of 4ml/hr. This epidural infusion will continue throughout the case. Titration of this infusion will be guided by clinical judgment of the primary anesthesia team in the operating room between the range of 0-14 ml/hr with primary assessments including the patient's analgesic requirement and hemodynamic stability.

Intraoperative period: A standardized anesthesia induction and maintenance protocol will be used. This protocol will include sedation with 2mg of midazolam and fentanyl (1-2mcg/kg) for epidural placement, 2-3 μg/kg fentanyl prior to induction, 2-2.5mg/kg propofol on induction and isoflurane for maintenance of anesthesia. Additional narcotic administration is at the discretion of the primary anesthesia team but recommended for patients up to their daily opiate dose, plus an additional 0.1mg/kg morphine at or before emergence. Ketorolac 15mg may be administered as clinically indicated unless contraindications such as age >75, renal insufficiency (gfr <60) or surgeon preference. In addition, 4mg dexamethasone will be administered on induction. Nitrous oxide and ketamine will not be used. Hemodynamic monitoring will be accomplished with standard monitors, an arterial line placed by the primary anesthesia team, and, if indicated, noninvasive cardiac outcome monitors. The arterial line will be placed according to the preference of the primary anesthesia team.

Postoperative period: Post operative pain management will be dictated by the primary surgical service. Typical management includes patient-controlled analgesia of IV morphine, fentanyl or hydromorphone with transition to oral medications as indicated on post operative day one. Titration of the epidural between the 4cc/hr up to a maximum of 14cc/hr will be made based upon a specific protocol for inadequate pain relief. The epidural will be bolused with 4cc from the standard solution and then the rate of the infusion will be increased by 2cc/hr if and when a patient requires better analgesia. If the epidural is deemed non functioning by the supervising attending on the pain service, as evidence by a lack of sensory blockade in the distribution of the incision and patient discomfort, then it is at the discretion of the acute pain service attending to remove or replace the non-functional epidural.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for open thoracotomy procedure
* Patient provides informed consent

Exclusion Criteria:

* Age less than 19
* Pregnancy
* Contraindication to an epidural catheter placement bleeding disorder cardiac valve stenosis systemic infection spinal abnormality
* Allergy to local anesthetics or X-ray dye
* Patient refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parra MC, Washburn K, Brown JR, Beach ML, Yeager MP, Barr P, Bonham K, Lamb K, Loftus RW. Fluoroscopic Guidance Increases the Incidence of Thoracic Epidural Catheter Placement Within the Epidural Space: A Randomized Trial. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):17-24. doi: 10.1097/AAP.0000000000000519. PMID 27922948

RESULTS

PARTICIPANT FLOW:
Groups:
- Traditional: The traditional approach for placement of an epidural catheter is indirect indicators of placement including palpation of spine and 'loss-of-resistance' to fluid injection.
  Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr into the epidural catheter for pain control.
  Traditional: An epidural catheter is placed before surgery with the patient sitting. The catheter is placed using indirect indicators of placement: depth of needle and ability to inject solution through the needle ('loss of resistance'). After needle placement in the epidural space, an epidural catheter is threaded through the needle and the needle removed. After catheter is placed, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected to exclude intravascular placement. A continuous infusion of 1/8% bupivacaine is started at 4ml/hr. The bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusion rate by 2ml/hr up to a maximum of 14ml/hr.
- Fluoroscopy: Real-time fluoroscopic X-ray guidance to confirm placement of an epidural catheter in the epidural space at the desired location.
  Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr during and after surgery for pain control.
  Fluoroscopy: Device: Fluoroscopy Patients lie prone on X-ray compatible operating table and an X-ray device obtains X-ray images of catheter placement. An epidural catheter is placed with local anesthesia as a needle that is advanced into the epidural space. A catheter is then placed through the needle to the desired location and the needle is removed. After the catheter is placed, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected into the catheter to exclude intravascular placement. Following this, a continuous infusion of 1/8% bupivacaine is started at 4ml/hr. The bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusion rate by 2ml/hr up to a maximum of 14ml/hr
Period: Overall Study
Arm/Group | Traditional | Fluoroscopy
Started | 53 | 47
Completed | 53 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluoroscopy: Real-time fluoroscopic X-ray guidance to confirm placement of epidural catheter in the epidural space at the desired location.
  Following epidural catheter placement 1/8% bupivacaine is infused at 4ml/hr during and after surgery for pain control.
  Fluoroscopy: Device: Fluoroscopy Patients lie prone on X-ray compatible operating table and an X-ray device obtains images of epidural catheter placement. An epidural catheter is placed with local anesthesia as a needle that is advanced into the epidural space. A catheter is then placed through the needle to the desired location and the needle is removed. After the catheter is placed, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected into the catheter to exclude intravascular placement. Following this, a continuous infusion of 1/8% bupivacaine is started at 4ml/hr. After surgery, the bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusion rate by 2ml/hr up to a maximum of 14ml/hr
- Traditional: The traditional approach for placement of an epidural catheter is with indirect indicators including palpation of spine and 'loss-of-resistance' to fluid injection.
  Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr during and after surgery for pain control.
  Traditional: An epidural catheter is placed before surgery with the patient sitting. The catheter is placed using indirect indicators of proper placement: depth of needle insertion and ability to inject solution through the needle ('loss of resistance'). After needle placement, an epidural catheter is threaded through the needle and the needle removed. After catheter is placement, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected to exclude intravascular placement. A continuous infusion of 1/8% bupivacaine is started at 4ml/hr. After surgery, the bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusion rate by 2ml/hr up to a maximum of 14ml/hr.
- Total: Total of all reporting groups
Arm/Group | Fluoroscopy | Traditional | Total
Number analyzed (Participants) | 47 | 53 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 34 | 59
  >=65 years | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (10.6) | 64.9 (8.9) | 65.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 51
  Male | 25 | 24 | 49
Region of Enrollment [Number; unit: participants]
  United States | 47 | 53 | 100

OUTCOME MEASURES:

1. Primary Outcome: Intravenous Pain Medication
Description: Outcome measure is mg of morphine equivalent used in first 24 hours after surgery: Postoperative pain medication use during the first 24 postoperative hours will be calculated by converting medication to an equivalent amount of morphine. This is an indirect measure of postoperative pain.
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: milligrams
Groups:
- Fluoroscopy: Real-time fluoroscopic X-ray guidance to confirm placement of an epidural catheter.
  Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr into the epidural catheter during and after surgery for pain control.
  Fluoroscopy: Device: Fluoroscopy Patients lie prone on X-ray compatible operating table and an X-ray device obtains X-ray images of epidural catheter placement. An epidural catheter is placed with local anesthesia as a needle that is advanced into the epidural space. A catheter is then placed through the needle to the desired location and the needle is removed. After the catheter is placed, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected into the catheter to exclude intravascular placement. Following this, a continuous infusion of 1/8% bupivacaine is started at 4ml/hr. After surgery, the bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusi
- Traditional: The traditional approach for placement of an epidural catheter is used with indirect indicators of placement including palpation of spine and 'loss-of-resistance' to fluid injection.
  Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr into the epidural catheter during and after surgery for pain control.
  Traditional:An epidural catheter is placed before surgery with the patient sitting at bedside. The catheter is placed with local anesthesia using indirect indicators of proper placement: depth of needle insertion and ability to inject solution through the needle ('loss of resistance'). After needle placement in the epidural space, an epidural catheter is threaded through the needle 3-4 cm and the needle removed. After catheter is placement, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected into the catheter to exclude intravascular placement. Following this, a continuous infusion of 1/8% bupivacaine is started at 4ml/hr. After surgery, the b
Arm/Group | Fluoroscopy | Traditional
Number analyzed (Participants) | 47 | 53
milligrams | 63 (33) | 66 (27)

2. Secondary Outcome: Incidence of Epidural Catheter Failure
Description: Percent of epidural catheters that were correctly placed (percentage of catheters).
Time Frame: 24 hours after surgery
Measure: Number; unit: percentage of catheters
Arm/Group | Fluoroscopy | Traditional
Number analyzed (Participants) | 47 | 53
percentage of catheters | 74 | 98

3. Secondary Outcome: Postoperative Pain Intensity Measured by Numeric Scale
Description: Assessment of pain intensity by verbal report of patient on a digital scale of 0 (no pain) to 10 (worst pain).
Time Frame: Measured at 24 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale of 0 to 10
Arm/Group | Fluoroscopy | Traditional
Number analyzed (Participants) | 47 | 53
units on a scale of 0 to 10 | 6.3 (3.1) | 6.6 (3.4)

4. Secondary Outcome: Postoperative Pain Intensity Measured by Numeric Scale
Description: Assessment of pain intensity by verbal report of patient on a digital scale of 0 (no pain) to 10 (worst pain).
Time Frame: Measured at 48 hours after surgery
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Fluoroscopy | Traditional
Number analyzed (Participants) | 47 | 53
milligrams | 6.4 (3.3) | 6.8 (2.7)

5. Secondary Outcome: Postoperative Pain Intensity Measured by Numeric Scale
Description: Assessment of pain intensity by verbal report of patient on a digital scale of 0 (no pain) to 10 (worst pain).
Time Frame: 3 months after surgery during follow up office visit with surgeon
Population: Insufficient data were collected for this analysis
Arm/Group | Fluoroscopy | Traditional
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Fluoroscopy: Real-time fluoroscopic X-ray guidance to confirm placement of an epidural catheter Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr during and after surgery for pain control.
  Fluoroscopy: Device: Fluoroscopy Patients lie prone on X-ray compatible operating table and an X-ray device obtains X-ray images of epidural catheter placement. An epidural catheter is placed with local anesthesia as a needle that is advanced into the epidural space. A catheter is then placed through the needle to the desired location and the needle is removed. After the catheter is placed, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected into the catheter to exclude intravascular placement. Following this, a continuous infusion of 1/8% bupivacaine is started at 4ml/hr. After surgery, the bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusion rate by 2ml/hr up to a maximum of 14ml/hr
- Traditional: The traditional approach for placement of an epidural catheter is used with indirect indicators of placement.
  Following epidural catheter placement, 1/8% bupivacaine is infused at 4ml/hr during and after surgery for pain control.
  Traditional: An epidural catheter is placed before surgery with the patient sitting at bedside. The catheter is placed with local anesthesia using indirect indicators of proper placement: depth of needle insertion and ability to inject solution through the needle ('loss of resistance'). After needle placement, an epidural catheter is threaded through the needle and the needle removed. After catheter is placement, a test dose of 1.5% lidocaine with 5ug/cc epinephrine is injected into the catheter to exclude intravascular placement. Following this, a continuous infusion of 1/8% bupivacaine is started at 4ml/hr. After surgery, the bupivacaine infusion may be adjusted with bolus injections of 2ml and/or increase in the infusion rate by 2ml/hr .
Arm/Group | Fluoroscopy | Traditional
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/53
Other Adverse Events (participants affected / at risk) | 0/47 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No